CLINICAL TRIAL: NCT06137118
Title: A Phase 1/2 Study to Evaluate the Safety and Efficacy of AZD0486 in Adolescent and Adult Participants With Relapsed or Refractory B-Cell Acute Lymphoblastic Leukaemia
Brief Title: AZD0486 as Monotherapy in B-cell Acute Lymphoblastic Leukaemia
Acronym: SYRUS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7405C00001
Record Dates: First submitted 2023-11-03; First posted 2023-11-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: B-cell Acute Lymphoblastic Leukemia (B-ALL)
Keywords: B-cell acute lymphoblastic leukemia; Leukemia; B-lymphocytes; AZD0486
MeSH Terms: conditions — Burkitt Lymphoma; Leukemia

STUDY DESIGN:
Intervention Model Description: The trial will assess AZD0486 IV infusion in monotherapy. Part A will evaluate ascending dose levels of AZD0486 in participants 12 years and above with B-ALL. Part B will evaluate up to 2 safe-declared dose levels in participants with both Ph(+) and Ph(-) B-ALL aged 12 years and above to select the RP2D. Part C will expand the RP2D dose level cohort to assess efficacy in a large number of subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: AZD0486 Dose Escalation (Experimental): Ascending dose level cohorts of AZD0486 in B-ALL participants aged 12 years and above.
  Interventions: Drug: AZD0486
- Part B: Dose Optimization (Experimental): Up to 2 cohorts will be evaluated prior declared safe-doses and schedules in order to determine the recommended phase 2 dose (RP2D). Participants, aged 12 years and above, will receive AZD0486 IV infusions and will be randomized in a 1:1 ratio.
  Interventions: Drug: AZD0486
- Part C: Dose Expansion (Experimental): Part C will consist of 1 cohort of participants aged 12 years and above, treated with the optimal dose selected in Part B and receive IV AZD0486 monotherapy.
  Interventions: Drug: AZD0486

INTERVENTIONS:
Drug: AZD0486 — Investigational Product administered via intravenous infusion.

SUMMARY:
This is a Phase 1/2, global multicentre, open-label, single-arm, dose escalation and dose optimisation study of AZD0486 to evaluate the safety, tolerability, and efficacy of AZD0486 monotherapy in participants with R/R B ALL who have received ≥ 2 prior lines of therapies. The study will consist of 3 parts. Part A monotherapy dose escalation. Part B dose optimisation. Part C Dose expansion at the recommended phase 2 dose (RP2D)

DETAILED DESCRIPTION:
This dose escalation and optimization study is evaluating the safety, tolerability, PK, PD and clinical activity of AZD0486 monotherapy in r/r B-ALL.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12 years and above (Parts A, B and C).
* Participants with B-cell Acute Lymphoblastic Leukemia with CD19 expression by local lab with:

  1. Bone marrow infiltration with >/= 5% blasts
  2. Either relapsed or refractory after a minimum of 2 prior therapies or after 1 prior line of therapy if no SOC available option.
  3. Philadelphia positive participants are allowed in all parts of the study, if intolerant or refractory to TKIs.
* For participants older than 16 years, Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 2. For Participants 16 years or younger, Lansky score more or equal to 50%.

The above is a summary, other inclusion criteria details may apply.

Exclusion Criteria:

* Active CNS involvement by B-ALL, defined by presence of ALL blasts in CSF (CNS2 and CNS3 criteria).
* Isolated extramedullary disease relapse.
* Testicular leukemia
* History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis; or prior Grade 4 neurotoxicity with CAR-T or TCE therapy.
* History of other malignancy (with certain exceptions).
* Unresolved AEs >/= Grade 2, from prior therapies
* Prior therapy with TCEs within 4 weeks, CAR T-cell therapy or autologous HSCT within 8 weeks or prior alloSCT within 12 weeks of start of therapy.
* GVHD requiring immunosuppressive therapy within 3 weeks prior to AZD0486 treatment.

The above is a summary, other exclusion criteria details may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2026-11-13 (Estimated); Study Completion 2027-06-29 (Estimated)

PRIMARY OUTCOMES:
Part A: Frequency of DLTs | Up to 28 days
  DLTs are dose-limiting toxicities as defined in the study protocol
Parts A & B: Safety Evaluation of AZD0486 | From signing of informed consent through data cutoff, up to 42 months
  Frequency, severity, and relationship to study drug of AEs and SAEs; dose modifications; changes in laboratory evaluations; QTc, and vital signs changes.
Parts B & C: Rate of CR within 3 cycles | Up to three cycles of 28 days each
  To evaluate the efficacy of AZD0486 based on NCCN response criteria (in Part B and C).

SECONDARY OUTCOMES:
Part A: Rate of CR within 3 cycles | Up to 3 cycles of 28 days each
  the percentage of participants with a best response of CR within 3 cycles based on NCCN response criteria by investigators
Part A,B,C: Rate of CR/CRh and CR/CRh/CRi within 3 cycles | Up to 3 cycles of 28 days each
  proportion of participants achieving CR/CRh/CRi within 3 cycles based on NCCN response criteria by investigators (Part A) based on the response evaluable population, and by central review confirmation (Parts B and C) based on the FAS.
Parts A, B, C: Rate of CR, CR/CRh and CR/CRh/CRi at any time during the study | From first dose to end of treatment or data cutoff, whichever comes first, assessed up to 42 months
  Rate of CR, CR/CRh and CR/CRh/CRi at any time during study (Best CR, best CR/CRh and best CR/CRh/CRi)
Parts A, B, C: Duration of CR, CR/CRh and CR/CRh/CRi | From first dose to last progression or data cutoff, whichever comes first, assessed up to 42 months
  the time from the date of first documented CR, CR/CRh, or CR/CRh/CRi response, respectively, until the date of documented relapse or death due to any cause in the absence of disease progression or relapse, whichever occurs earlier.
Parts A, B, C: Event-free survival (EFS) | From First dose to last progression or data cutoff, whichever comes first, assessed up to 42 months
  Event-free survival is defined as the time from the date of the first dose until the date of a relapse after achieving a CR/CRh/CRi, or death due to any cause, whichever occurs first.
Parts A, B, C: Overall Survival (OS) | From First dose to data cutoff, up to 42 months
  The OS is defined as the time from date of first dose until death due to any cause regardless of whether the participant withdraws from treatment or receives a TTNT.
Parts B &C: Subsequent alloSCT or donor lymphocyte infusion if used as an alloSCT substitute | From first dose to EOT, up to 42 Months
  Percentage of participants who received a subsequent alloSCT, or DLI if used as an alloSCT substitute, post AZD0486 treatment
Part A, B, C:MRD-negative rate of CR | From First dose to data cutoff, up to 42 months
  To evaluate the impact of AZD0486 on MRD-negative rate of CR, CR/CRh and CR/CRi
Parts A, B, & C: PK characterization of AZD0486 | From first dose to data cutoff, up to 42 months
  Derived PK parameter: AUC
Parts A, B & C: PK Characterization of AZD0486 | From first dose to data cutoff, up to 42 months
  Derived PK parameter: Cmax
Parts A, B, C: PK Characterization of AZD0486 | From first dose to data cutoff, up to 42 months
  Derived PK Parameter: tmax
Parts A, B, C: PK Characterization of AZD0486 | From first dose to data cutoff, up to 42 months
  Derived PK parameter: Ctrough
Parts A, B, C: PK Characterization of AZD0486 | From first dose to data cutoff, up to 42 months
  Derived PK Parameter: t1/2
Parts A, B, C: PK Characterization of AZD0486 | From first dose to data cutoff, up to 42 months
  Derived PK Parameter: CL of AZD0486
Parts A, B, C: ADA characterization of AZD0486 | From First dose to EOT, up to 42 months
  Summary of pre-existing and treatment-induced ADAs for AZD0486 (positive or negative, titres)
Part C: Safety Evaluation of AZD0486 | From signing of informed consent through completion of study treatment, an average of 6 months
  Frequency, severity, and relationship to study drug of AEs and SAEs; dose modifications; changes in laboratory evaluations; QTc, and vital signs changes.

CONTACTS AND LOCATIONS:
Locations (70):
- United States (12):
  - Research Site, Birmingham, Alabama
  - Research Site, Duarte, California
  - Research Site, Los Angeles, California
  - Research Site, Palo Alto, California
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, New York, New York
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin
- Research Site, Melbourne, Australia
- Brazil (2):
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (8):
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Nanjing
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Zhengzhou
- France (6):
  - Research Site, Caen
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Toulouse
- Germany (10):
  - Research Site, Cologne
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, München
  - Research Site, Münster
  - Research Site, Würzburg
- Italy (5):
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Roma
- Japan (11):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Kashiwa
  - Research Site, Kyoto
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Toyohashi
  - Research Site, Yamagata
- Research Site, Seoul, South Korea
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Salamanca
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (3):
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home